CLINICAL TRIAL: NCT06576570
Title: Evaluation and Modification of Surgeon Ergonomics in the Operation Room Using Artificial Intelligence Analytics
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB202301655
Record Dates: First submitted 2024-08-21; First posted 2024-08-28 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Work Related Upper Limb Disorder; Musculoskeletal Pain
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Intervention Model Description: Within-subject pre-post design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acute Care Surgery Attending and Resident Surgeons (Other): Participants will be asked to perform their normal operative work for 5 cases while being filmed. Data will be collected using the SoterTask™ software which calculates momentary data on risk and an aggregate risk level. Two standard ergonomic risk assessments: Rapid Upper Limb Assessment (RULA) or the Rapid Entire Body Assessment (REBA) are also calculated. Both assessments are current best practice standard for determining the level of ergonomic risk. The RULA and REBA data calculated by SoterTask will be compared to scores assessed by the research team from the same video recordings of the work tasks.
  Following the fifth operative case, participants will view an educational presentation of surgical ergonomics and review the data summarized from the ergonomic measurement system with video of their movement with a visual guideline highlighting high-risk angles and movements including legs, arms, neck and back.
  Interventions: Behavioral: Education presentation of surgical ergonomics; Behavioral: Summary of Ergonomic Measurement System

INTERVENTIONS:
Behavioral: Education presentation of surgical ergonomics — During an individual meeting with participant, a brief presentation will be supplied for review.
Behavioral: Summary of Ergonomic Measurement System — Participant will view a video of their movements with a visual guideline highlighting high-risk angles and movements.

SUMMARY:
The study is working to identify actions of surgeons in the operating room that can contribute to work-related musculoskeletal disorders. This includes poor positioning and time spent in poor positioning while working in the operating room. The study is also looking to determine if fatigue plays a role in work-related musculoskeletal disorders and whether an education intervention will change ergonomic risk.

DETAILED DESCRIPTION:
The study is working to identify actions of surgeons in the operating room that can contribute to work-related musculoskeletal disorders. This includes poor positioning and time spent in poor positioning while working in the operating room. The study is also looking to determine if fatigue plays a role in work-related musculoskeletal disorders.

Employing within-subject pre-post design to assess 1) patterns of aggregate risk data from video analysis in the OR for resident and attending surgeons over time and for different types of surgical tasks, 2) concurrent reliability assessment of the Rapid Upper Limb Assessment and Rapid Entire Body Assessment scores calculated from the software and visual analysis, 3) changes in pain data after review of the SOTER Task ergonomic outputs. The feasibility of using the system in the OR will also be assessed for open and laparoscopic surgery.

The study team will collect data, perform assessments, collect information from self-proctored surveys, and video record surgeon activities in the operating room on 20 surgeons. The video recordings will take measurements to assess risk factors for work-related musculoskeletal disorders. Following the fifth surgical case, the study team complete an education intervention by reviewing measurements established in the video recordings and supply a brief presentation on Ergonomics for Surgeons. A summary of observed body positioning for each subject is provided. Post intervention, five additional surgical cases will be observed in the manner of the previous cases to identify change in ergonomic risk.

ELIGIBILITY:
Inclusion Criteria:

• Any general surgery operative case by a surgeon from the Division of Acute Care Surgery. These cases will be conducted in what has been designated as the "Acute Care Surgery OR" for the day.

Exclusion Criteria:

* Any operative case in which the surgical attending or resident has not signed informed consent to record this individual during the case.
* Any operative case that the surgical attending feels is inappropriate for video recording or when filming could interfere with surgical procedures

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2026-10-15 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Determine Ergonomic Risk Through Video-based Analysis calculated by an artificial intelligence software and evaluator assessment of Rapid Upper Limb Assessment (RULA) and Rapid Entire Body Assessment (REBA) | 1 year
  determine the ergonomic risk experienced by surgical attendings and residents during open and laparoscopic surgery measured through video-based analysis of

SECONDARY OUTCOMES:
Change in Ergonomic Risk After Reviewing Video Capture and Risk Data | 1 year
  determine if there is any change in ergonomic risk after reviewing video capture and risk data collated through artificial intelligence algorithms

CONTACTS AND LOCATIONS:
Overall Officials: Philip Efron, MD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - UF Health at Shands Hospital, Gainesville, Florida
  - UF Health Shands Hospital at the University of Florida, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: No